CLINICAL TRIAL: NCT06679647
Title: Acceptability, Usability and Preliminary Effectiveness of ChatGPT in Increasing Seasonal Influenza Vaccination Uptake Among Older Adults in Hong Kong
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SIV_ChatGPT
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Behavior Change Interventions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ChatGPT group (Experimental): Participants will be invited to use a trained ChatGPT which answers questions related to seasonal influenza vaccination. The functions can be used repeatedly throughout the intervention period (4 weeks), and participants will be free to spend as much time as they want on such functions.
  Interventions: Behavioral: Access to a trained ChatGPT

INTERVENTIONS:
Behavioral: Access to a trained ChatGPT — Participants will be invited to use a trained ChatGPT which answers questions related to seasonal influenza vaccination. The functions can be used repeatedly throughout the intervention period (4 weeks), and participants will be free to spend as much time as they want on such functions.

SUMMARY:
In this project, we will train a ChatGPT to provide real-time answers to questions related to the SIV for older adults in Hong Kong.

This study aims to evaluate the usability, acceptability, and preliminary effectiveness of the ChatGPT among 50 community-living people aged 65 years and above in Hong Kong.

The primary objectives are to evaluate the usability and acceptability (including the extent of usage and subjective experiences of behavioural, cognitive, and affective engagement) of the ChatGPT at the end of the 4-week intervention period (T1).

The secondary objectives are to evaluate the following conditions measured at T1, as compared to those measured at baseline (T0):

1. Self-reported uptake of SIV in the past month.
2. Changes in behavioural intention to receive SIV for the approaching flu season.
3. Changes in knowledge and attitudes related to SIV.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years;
* Possession of a Hong Kong ID;
* Able to speak and comprehend Cantonese;
* Have a smartphone with internet access;
* Have not taken SIV for the approaching flu season.

Exclusion Criteria:

* With diagnosis of cognitive impairment or dementia;
* Either blindness or deafness;
* With known contraindications to the SIV as indicated by the Hong Kong Centre for Health Protection

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Perceived usability | 1 month
  Perceived usability assessed by the validated Chinese version of the 10-item Perceived Usability Scale (SUS)
Extent of usage documented by the ChatGPT | 1 month
  Extent of usage documented by the ChatGPT
Subjective experiences related to behavioural, cognitive, and affective engagement | 1 month
  Subjective experiences related to behavioural, cognitive, and affective engagement measured by the validated Twente Engagement with eHealth Technologies Scale (TWEETS)

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, PhD, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Z, Tsang TH, Yu FY, Fang Y, Chen S, Sun F, Mo PKH, Wong KC. Effectiveness, Usability, and Acceptability of ChatGPT With Retrieval-Augmented Generation (SIV-ChatGPT) in Increasing Seasonal Influenza Vaccination Uptake Among Older Adults: Quasi-Experimental Study. J Med Internet Res. 2025 Sep 8;27:e76849. doi: 10.2196/76849. PMID 40921067